CLINICAL TRIAL: NCT03944460
Title: A Randomized, Double-blind and Placebo-controlled Single Ascending-dose Phase I Study (First-in-human) to Investigate the Safety, Tolerability and Pharmacokinetics of Contraloid Acetate (in Healthy Subjects).
Brief Title: SAD Phase I Study (First-in-human) to Investigate Contraloid Acetate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prof. Dr. Dieter Willbold (Other)
Collaborators: Helmholtz-Gemeinschaft Deutscher Forschungszentren, Germany (Unknown); Medical University of Vienna (Other); NeuroScios, Austria (Unknown); Triskelion, The Netherlands (Unknown); Fundación Teófilo Hernando, Spain (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Dieter Willbold, Director of Institute of Complex Systems, Structural Biochemistry (ICS-6), Forschungszentrum Juelich
Organization: Forschungszentrum Juelich (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EUDRA-CT: 2017-000396-93
Record Dates: First submitted 2019-04-26; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer Dementia; Alzheimer Disease
Keywords: anti-prionic; anti-Abeta-pionic; treatment of cognition and memory deficits; AD patients; AD stage-independent; NOT anti-amyloid; neuron specific Ca-ion reduction
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multi-cohort trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Contraloid 4 mg (Active Comparator): 4 mg Contraloid/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Contraloid 12 mg (Active Comparator): 12 mg Contraloid/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Contraloid 36 mg (Active Comparator): 36 mg Contraloid/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Contraloid 108 mg (Active Comparator): 108 mg Contraloid/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Contraloid 320 mg (Active Comparator): 320 mg Contraloid/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Placebo (for Contraloid) 4 mg (Placebo Comparator): 4 mg placebo/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Placebo (for Contraloid) 12 mg (Placebo Comparator): 12 mg placebo/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Placebo (for Contraloid) 36 mg (Placebo Comparator): 36 mg placebo/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Placebo (for Contraloid) 108 mg (Placebo Comparator): 108 mg placebo/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid
- Placebo (for Contraloid) 320 mg (Placebo Comparator): 320 mg placebo/participant in a single oral dose with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Drug: Contraloid

INTERVENTIONS:
Drug: Contraloid — Oral administration of capsules, drug substance or placebo without any excipients.
  Other Names: PRI-002

SUMMARY:
This is a single-center first-in-human single-ascending-dose clinical trial assessing the safety and tolerability of oral dosing of Contraloid acetate in healthy volunteers. The study drug Contraloid (alias RD2, alias PRI-002) is an orally available all-D-peptide, which was developed to directly destroy toxic and replicating A-beta oligomer prions, by disassembling them into A-beta monomers. The study drug is specifically designed for the curative or at least disease-modifying treatment of cognition, memory and behavior deficits in Alzheimer´s disease patients. The study drug is not designed to reduce brain plaque load or total A-beta in cerebrospinal fluid. The study drug is blood-brain-barrier penetrable [1] and has demonstrated target engagement in vitro and in vivo [2, 3]. Preclinical treatments in three different transgenic mouse models in three different laboratories yielded improved cognition and deceleration of neurodegeneration, even under truly non-preventive treatment conditions and even when applied orally [2-5]. The hereby obtained PRI-002 plasma levels have also been achieved in humans after single oral dosing.

DETAILED DESCRIPTION:
The investigation on the compound Contraloid acetate in a single-ascending-dose phase I study (first-in-human) has been performed in 40 healthy male participants, randomly assigned to the treatment. Main focus was on the evaluation of the outcome of the safety and tolerability; secondarily the pharmacokinetic characteristics of the compound were assessed. Five different ascending doses (4, 12, 36, 108, and 320 mg Contraloid) administered orally as a single dose, were tested in five cohorts on respectively six participants per cohort, additionally two participants of each cohort received placebo.

In order to maintain the highest level of security for the participants of this first-in-human study a staggered design was used. First, only two sentinels of each cohort were administered with the study drug or placebo (ratio 1:1). Only after assessing all available data by the data safety and monitoring board (DSMB), the rest of the cohort (5 study drug : 1 placebo) were allowed to be treated. This took place on two consecutive days, administering the study drug to three participants per each starting day. After DSMB permission the next higher dose level was started in the next cohort with the same scheme of administration.

During the screening period the informed consent was obtained and the evaluation of the inclusion and exclusion criteria, collection of demographic data and previous medical history, physical examination and health assessment, 12-lead ECG were performed. Additionally vital signs, haemogram, coagulation, biochemistry and urine analysis determination, as well as serology and testing of drug abuse were carried out.

On the first study day the participants received in fasting conditions the study drug after re-evaluation the inclusion/exclusion criteria. For monitoring the laboratory parameters and the pharmacokinetics of Contraloid blood draws were performed in a predetermined frequency. Physical conditions, vital signs, ECG and EEG, concomitant medication, adverse events were monitored closely. Sentinels stayed in the Phase-I Unit for 72 hours, and the remaining participants of the cohort for 24 hours. A follow-up was performed on Days 3, 4 and 8. The study was double-blinded and conducted under the EU regulations and Good Clinical Practice (GCP) and national Austrian law. Monitoring and PV was performed by the CRO NeuroScios, DM by Fundación Teófilo Hernando, Spain, bio-analytics by Triskelion, The Netherlands.

Contraloid (alias RD2, alias PRI-002) is an all-D-peptide, which was developed to directly destroy toxic and replicating A-beta oligomer prions by disassembling them into A-beta monomers. The study drug is specifically designed for the curative or at least disease-modifying treatment of cognition, memory and behavior deficits in Alzheimer´s disease patients. The study drug is not designed to reduce brain plaque load or total A-beta in cerebrospinal fluid. The study drug is blood-brain-barrier penetrable [1] and has demonstrated target engagement in vitro and in vivo [2, 3]. Preclinical treatments in three different transgenic mouse models in three different laboratories yielded improved cognition and deceleration of neurodegeneration, even under truly non-preventive treatment conditions and even when applied orally [2-5]. The hereby obtained PRI-002 plasma levels have also been achieved in humans after single oral dosing.

ELIGIBILITY:
Inclusion Criteria:

* With clinical history and physical examination results within normality.
* Electrocardiogram without clinically significant pathologic abnormalities and with QTc values lesser than 450 ms.
* Normotensive as defined by Systolic Blood Pressure ≤ 150 mm Hg. Diastolic Blood Pressure ≤ 90 mm Hg.
* BMI between 19.0 and 30.0 kg/m2.
* Body weight between 55 and 85 kg, inclusive
* Signed ICF

Exclusion Criteria:

* Any chronic medical condition (such as type 1 diabetes) requiring chronic treatment that might increase the risk to the subject or confound the interpretation of safety observations.
* Evidence of active infection requiring antibiotic therapy within 14 days prior to screening.
* Medical history of vasculitis or any autoimmune disease excluding seasonal allergic rhinitis and childhood history of atopic dermatitis.
* History of any treatment for cancer within the past 2 years, other than basal cell or squamous cell carcinoma of the skin.
* Seropositive for human immunodeficiency virus (HIV).
* History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for Hepatitis B surface antigen [HbsAg] or anti-Hepatitis C [HCV] antibody).
* Clinically significant abnormalities in screening laboratory tests, including:

  * Absolute neutrophil count < 1.4 x109
  * Alanine transaminase (ALT) or aspartate transaminase (AST) > 1.5 x the upper limit of normal (ULN)
  * Absolute lymphocyte count < 1.2 x 109
  * Lactate dehydrogenase (LDH) > 1.5 x ULN
  * Total bilirubin level: Out of normal range 0-1.5 mg/dL
  * eGFR < 60 mL/min
  * Hemoglobin (Hgb): out of normal range (male: 13,5-18,0 g/dL)
  * CK level higher than normal values (250U/L)
* All prescription, over-the-counter and herbal medications are prohibited within 10 days prior to study dosing (with exception of calcium/vitamin D supplements, nasal steroids, ocular medications, and paracetamol ≤1000 mg/day at the discretion of the Investigator).
* Use of an investigational drug within 2 months prior to dosing in this study.
* Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs (e.g. small bowel disease, Crohn's disease, celiac disease, or liver disease.)
* Psychiatric history of current or past psychosis, bi-polar disorder, clinical depression, or anxiety disorder requiring chronic medication within the past 5 years.
* History of substance abuse, including alcohol
* Smokers
* History of substance or drug dependence, or positive urine drug screen at screening visit.
* History of head injury.
* Chronic kidney disease (defined as the presence of any degree of proteinuria on urine analysis and/or an eGFR of <60 ml/min using the MDRD formula).
* Any reason or opinion of the investigator that would prevent the subject from participation in the study.
* Inability to follow the instructions or an unwillingness to collaborate during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of Contraloid by monitoring vital signs, ECG, EEG, and lab values | 8 days
  To evaluate the safety and tolerability of Contraloid acetate in healthy subjects by assessing the number, severity and type of adverse events, including changes in vital signs, physical examinations, laboratory safety tests and ECGs.
Assessment of pharmacokinetics of Contraloid: Area under curve (AUC) in plasma | 72 hours
  Area under curve (AUC) in plasma
Assessment of pharmacokinetics of Contraloid: Cmax in plasma | 72 hours
  Cmax in plasma
Assessment of pharmacokinetics of Contraloid: Tmax in plasma | 72 hours
  Tmax in plasma
Assessment of pharmacokinetics of Contraloid: Terminal elimination half-life (t1/2) in plasma | 72 hours
  Terminal elimination half-life (t1/2) in plasma
Assessment of pharmacokinetics of Contraloid: Apparent total clearance (Cl/F) in plasma | 72 hours
  Apparent total clearance (Cl/F) in plasma
Assessment of pharmacokinetics of Contraloid: Volume of distribution (Vd) in plasma | 72 hours
  Volume of distribution (Vd) in plasma
AUC0-24 of Contraloid does not exceed of 2.3 µg·h/mL | 72 hours
  Additionally, the AUC0-24 values of Contraloid in plasma will be determined in order to ensure that the recommended AUC0-24 of Contraloid does not exceed of 2.3 µg·h/mL in any of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — University of Vienna
Locations (1):
- Forschungszentrum Jülich, Jülich, Germany

IPD SHARING:
Plan to Share IPD: No
Only as far as covered by the EU GDPR and regulated by GCP

REFERENCES:
- See also: Press releases of the research center Juelich — http://www.fz-juelich.de/ics/ics-6/EN/Home/home_node.html
- See also: Press releases of Priavoid — https://priavoid.com/